CLINICAL TRIAL: NCT05820451
Title: Impella Real-World Surveillance of Patients Using Sodium Bicarbonate
Status: Completed | Type: Observational
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ABMD-CIP-21-02-SS01
Record Dates: First submitted 2023-03-24; First posted 2023-04-19 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Cardiogenic Shock; High Risk PCI
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Left sided device: All patients implanted with a left sided support Impella device - this includes but is not limited to Impella 2.5, Impella CP, Impella 5.0, Impella 5.5.
  Interventions: Device: Impella CP, 2.5, 5.0 and 5.5 with Sodium Bicarbonate used as purge solution
- Right sided device: All patients implanted with a right sided support Impella device -this includes the Impella RP
  Interventions: Device: Impella RP with Sodium Bicarbonate used as purge solution

INTERVENTIONS:
Device: Impella CP, 2.5, 5.0 and 5.5 with Sodium Bicarbonate used as purge solution — US commercially approved Abiomed left sided hemodynamic support devices (Impella) will be included.
  Groups: Left sided device
Device: Impella RP with Sodium Bicarbonate used as purge solution — US commercially approved Abiomed right sided hemodynamic support devices (Impella) will be included.
  Groups: Right sided device

SUMMARY:
The population enrolled in this study are all subjects who received an Impella in which a bicarbonate-based purge solution was used.

ELIGIBILITY:
Left Sided Impella

Inclusion Criteria:

* Left-sided Impella with bicarbonate in the purge

Exclusion Criteria:

* Known LV thrombus

Right Sided Impella

Inclusion Criteria:

* Right-sided Impella with bicarbonate in the purge

Exclusion Criteria:

* Known pulmonary thromboemboli
* Known DVT

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects who received an Impella in which a bicarbonate-based purge solution was used
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint Left Sided Impella | From hospital admission until hospital discharge, average 5 days
  Rate of heiarchical composite of stroke, transient ischemic attack (TIA), left ventricular (LV) thrombus
Primary Endpoint Right Sided Impella | From hospital admission until hospital discharge, average 5 days
  Rate of heiarchical composite of pulmonary thromboemboli and deep vein thrombosis (DVT)

CONTACTS AND LOCATIONS:
Overall Officials: Amin Medjamia, MD, Study Director — Abiomed Inc.
Locations (20):
- United States (20):
  - University of Alabama, Birmingham, Alabama
  - Pima Heart and Vascular (Tuscon Medical Center), Tucson, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Keck USC Medical Center, Los Angeles, California
  - Advent Helath Orlando, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Henry Ford, Detroit, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Providence St. Patrick, Missoula, Montana
  - University of Nebraska, Omaha, Nebraska
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Christ Hospital, Cincinnatti, Ohio
  - Montefiore Medical Center - Moses, Portland, Oregon
  - Legacy Emanuel, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Baylor Scott and White (Baylor Heart and Vascular), Dallas, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Providence Sacred Heart, Spokane, Washington
  - MultiCare Tacoma General, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No